CLINICAL TRIAL: NCT01811654
Title: A Randomized, Pragmatic, Effectiveness Trial Evaluating Intra-articular Hyaluronan for the Symptomatic Treatment of Chronic Patellofemoral Pain Syndrome
Brief Title: Effectiveness Trial for Evaluating IAHA for PFPS
Acronym: PFPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-01020
Record Dates: First submitted 2013-02-15; First posted 2013-03-14 (Estimated); Results first posted 2020-02-13 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Patellofemoral; Hyaluronan; Intra-articular; Hyaluronic acid
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Viscosupplementation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Standard Care (No Intervention): Patients in this group will receive treatment per standard care. Standard Care is defined as consisting of physical therapy, activity modification (relative rest), and/or oral analgesic therapy. A specific physical therapy (PT) protocol will be implemented.
- Intra-Articular Hyaluronic Acid-Euflexxa (Active Comparator): Patients assigned to this group will receive treatment per standard care AND three (3) consecutive weekly injections of intra-articular hyaluronan (Euflexxa). Oral analgesics will be used at the lowest dose and for the shortest time possible to treat PFPS symptoms.
  Interventions: Device: Intra-Articular Hyaluronic Acid-Euflexxa

INTERVENTIONS:
Device: Intra-Articular Hyaluronic Acid-Euflexxa — IAHA was approved by the FDA in 1997 as a synovial fluid replacement device to help relieve the pain associated with knee osteoarthritis (OA) in patients who fail to respond adequately to conservative treatment and simple analgesics. In this study, IAHA, specifically Euflexxa, will be used off-label to determine whether patients afflicted with PFPS will experience similar analgesic effects as seen in those with OA.
  Other Names: Intra-articular Hyaluronan; IAHA; Viscosupplementation
  Arms: Intra-Articular Hyaluronic Acid-Euflexxa

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of intra-articular hyaluronan (IAHA) injections for the treatment of symptomatic patellofemoral pain syndrome (PFPS) and determine if this treatment can provide incremental clinical benefits over standard care for patients with this diagnosis.

DETAILED DESCRIPTION:
Objective: To determine the safety and effectiveness of intra-articular hyaluronan (IAHA) injections for the treatment of symptomatic patellofemoral pain syndrome (PFPS) and determine if this treatment can provide incremental clinical benefits over standard care for patients with this diagnosis.

Study Design: Two-arm, single-center, parallel, pragmatic, randomized, non-blinded, effectiveness trial

Indication for Use: For treatment of adult patients with Patellofemoral Pain Syndrome (PFPS) who have failed to respond to conservative treatment and simple analgesics (e.g. acetaminophen).

Setting: University Teaching Hospital, Faculty Practice

Subjects: Male and female patients aged 18-40 diagnosed with symptomatic patellofemoral pain syndrome (PFPS) that meet all inclusion and exclusion criteria. Approximately 68 subjects will be enrolled based on a power analysis of sample size estimation.

Methods: Patients signing informed consent will be randomized to one of two groups: (1) Standard Care, (2) Standard Care plus Intra-articular hyaluronan (IAHA) administered as a course of 3 consecutive weekly intra-articular injections.

Standard Care is defined as consisting of physical therapy, activity modification (relative rest), and/or oral analgesic therapy. Upon entering the trial, a specific physical therapy (PT) protocol will be implemented.

Data will be captured on the study knee history and symptoms. Radiographic examinations will be performed including weight-bearing anterior-posterior views with knees flexed 30 degrees, lateral, and sunrise views. The diagnosis of PFPS will be based on the subjects' being less than 40 years of age, and the occurrence of chronic retropatellar pain in the absence of other pain-causing abnormalities.

Arthrocentesis will be performed before all intra-articular injections, and any synovial fluid collected will be visually inspected for signs of infection before performing any injections. The volume of synovial fluid will be measured, and the samples will then be retained for further biomarker analysis.

A follow-up visit will be scheduled approximately 3 months after the baseline visit, to reevaluate patient condition.

Study Duration: A period of approximately 15 months is anticipated from the time the first patient is enrolled to the completion of the last patient visit. A final study report will then be generated after this 18 month time point.

ELIGIBILITY:
Inclusion Criteria:

* Adults from the ages of 18-40, male or female
* Diagnosis of unilateral OR bilateral patellofemoral pain syndrome
* Duration of diagnosis no less than 2 months and no greater than 3 years in the study knee
* Unresponsive to standard treatment of at least 6 weeks duration, consisting of physical therapy, activity modification (relative rest), and/or oral analgesic therapy
* Insidious onset of symptoms unrelated to a traumatic incident
* Pain described as "behind", "underneath", or "around" the patella reported during at least two of the following activities:

  * Going up or down stairs
  * Squatting
  * Running
  * Hopping or jumping
  * Kneeling
  * Prolonged sitting
* A baseline activity related VAS pain score between 50 and 90

Exclusion Criteria:

* Any co-morbidity that would influence the safety of intra-articular injections or impede safety and efficacy measurements in the study knee, such as:

  * Coagulopathies or the use of anticoagulant medications
  * History of allergy to any of the treatment interventions planned
  * Acute inflammation and/or palpable effusion in the study knee
  * Current or history of musculoskeletal infection in the study knee
  * Severe malalignment, deformity or chronic subluxation of study knee
  * History of prior patellar dislocation of the study knee
  * Ipsilateral joint/limb conditions (e.g. hip, thigh, lower leg, ankle, foot)
* Any condition other than PFPS in the contralateral knee present at the time of enrollment or developing during the course of enrollment
* Any radiographic signs of the following:

  * Osteoarthritis in any of the study knee compartments
  * Osteochondritis dissecans (OCD) lesions
  * Physeal injuries
  * Bone tumors
* Vulnerable subjects and pregnant women
* Participation in any other musculoskeletal studies

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2016-12-07 (Actual); Study Completion 2017-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Cardone, DO, Principal Investigator — NYU Langone Medical Center; Philip Band, PhD, Study Director — NYU Langone Medical Center/Hospital for Joint Disease
Locations (1):
- Center for Musculoskeletal Care - NYU Langone Medical Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Care | Intra-Articular Hyaluronic Acid-Euflexxa
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intra-Articular Hyaluronic Acid-Euflexxa | Standard Care | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 14 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 16 | 14 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Analog Scale (VAS) Score
Description: A 100mm visual analog scale (VAS) for activity related pain assessment will serve as the primary outcome measure. The 2-sample t-test comparing the two treatment groups' mean change from baseline issued. No pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm). The 2 sample t-test approximates the test of the null hypothesis that there is a difference in mean change from baseline in the VAS for activity-related pain between the HA group and control group. Higher scores indicate higher level of pain.
Time Frame: At baseline and 3 month follow-up
Population: Both " Overall Number of Participants Analyzed" and "Participant Flow" are now consistent
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Standard Care | Intra-Articular Hyaluronic Acid-Euflexxa
Number analyzed (Participants) | 14 | 16
millimeters
  Baseline | 70 (13.59) | 62.23 (15.48)
  3 Months | 37.61 (31.40) | 25.025 (15.5)

2. Secondary Outcome: PFPS Severity Scale (PSS) Score
Description: Encompasses 10 statements regarding PFPS pain. Severity scale consists of 10 statements, rated from "0" indicating "no pain" and a "10" indicating "pain as bad as it could be."
Time Frame: 3 month follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Care | Intra-Articular Hyaluronic Acid-Euflexxa
Number analyzed (Participants) | 14 | 16
score on a scale
  Climbing stairs | 5 (2.44) | 5.21 (2.32)
  squatting | 5.5 (3.46) | 4.42 (3.77)
  walking | 3.5 (2.22) | 3.64 (2.37)
  Jogging | 3.87 (4.08) | 3.42 (3.56)
  Running | 3.75 (4.37) | 4.07 (4.08)
  sport | 2.06 (3.76) | 3.64 (3.95)
  sitting with bent | 5.81 (2.71) | 4.35 (2.92)
  kneeling | 4.56 (3.66) | 5.21 (2.51)
  pain at rest | 4.06 (2.54) | 2.57 (2.10)
  following activities | 4.75 (3.06) | 4.42 (2.62)

ADVERSE EVENTS:
Arm/Group | Standard Care | Intra-Articular Hyaluronic Acid-Euflexxa
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 0/14 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes